CLINICAL TRIAL: NCT06941792
Title: Effectiveness of Inclisiran for Patients With Coronary Heart Disease in China: a Multicenter, Standard of Care-Controlled Pragmatic Randomized Trial
Brief Title: Inclisiran Effectiveness in China: a Pragmatic Randomized Trial
Acronym: V-INVINCIBLE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKJX839A1CN06
Record Dates: First submitted 2025-03-06; First posted 2025-04-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease
Keywords: Inclisiran; effectiveness; lipid-lowering; low-density lipoprotein cholesterol Test on Target
MeSH Terms: conditions — Coronary Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inclisiran group (Experimental): patients in the inclisiran group will receive inclisiran (may or may not plus cholesterol absorption inhibitor at the discretion of the treating physician).
  Interventions: Drug: inclisiran sodium injection
- Standard of Care group (Active Comparator): Patients in the SoC group will switch to/add on another/other LLT(s) at the discretion of the treating physician, as long as it is not inclisiran or an investigational drug.
  Interventions: Combination Product: Standard of Care

INTERVENTIONS:
Drug: inclisiran sodium injection — After randomization, patients in the inclisiran group will receive inclisiran sodium injection
  Arms: inclisiran group
Combination Product: Standard of Care — After randomization switching to or adding on another/other lipid-lowering therapies
  Arms: Standard of Care group

SUMMARY:
The current study will be conducted to evaluate the real-world effectiveness of inclisiran relative to standard of care (SoC) in Chinese patients with coronary heart disease (CHD), not only with the low-density lipoprotein cholesterol (LDL-C) change in 1 year, but also the LDL-C Test on Target for 1 year. This study further aims to assess the adherence, treatment patterns and satisfaction, and safety of inclisiran among Chinese patients.

DETAILED DESCRIPTION:
The study is a multicenter, randomized, parallel, open-label, pragmatic trial, to assess the effectiveness of inclisiran in the real-world compared to SoC, in patients with CHD in China who did not achieve LDL-C goal despite maximally tolerated statin therapy for ≥4weeks stable using. CHD patients include patients with acute coronary syndrome and patients with chronic coronary syndrome.

After granting informed consent, being screened, and confirmed eligible for the study, participants will be randomized to 2 arms (inclisiran or SoC) in a 1:1 ratio.

Following the randomization, participants start inclisiran or SoC adaptation (which means switching to or adding on another/other lipid-lowering therapies (LLT[s]). This start date is defined as Day 0.

During follow-up, each participant will follow routine care, and the results of LDL-C tests will be collected for each Visit (every 3 months), with an allowable window of ±1.5 months. Each patient will be followed up until his/her end of study (EOS), which is the earliest of the end of follow-up period (Visit 4: approximately 12 months following Day 0), lost to follow-up, consent withdrawal, death, and participating in another interventional trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Documented diagnosis of CHD prior to screening, including acute coronary syndrome (ACS) and chronic coronary syndrome (CCS)
3. Aged ≥18 years at randomization
4. Despite maximally tolerated statin therapy for ≥4weeks stable using prior to screening, LDL-C result at screening not at goal (≥1.8 mmol/L).

The maximum tolerated dose of statins also includes patients with statin intolerance or contraindication.

Exclusion Criteria:

1. Received inclisiran during the 2 years prior to the screening.
2. Received proprotein convertase subtilisin-kexin type 9 (PCSK9) mabs during the 3 months prior to screening.
3. Participating in an interventional trial at enrollment
4. Having severe liver disorder (Child-Pugh class C)
5. Any other condition that may put the participant at significant risk if the participant participate in the current study, according to investigator's (or delegate's) judgment.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1590 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The percentage change in low-density lipoprotein cholesterol (LDL-C) level from baseline at 12 months, for the inclisiran group versus the standard of care (SoC) group | 12 months
  To evaluate the real-world effectiveness of inclisiran, on the change in LDL-C levels at Month 12, compared with SoC, in Chinese patients with coronary heart disease (CHD)

SECONDARY OUTCOMES:
The proportion of participants with the 1-year LDL-C Test on Target ≥75%, for the inclisiran group versus the SoC group | 12 months
  To evaluate the real-world effectiveness of inclisiran, on the LDL-C Test on Target at Month 12, compared with SoC, in Chinese patients with CHD
The percentage change in LDL-C level from baseline at 3 months, 6 months, and 9 months, for the inclisiran group versus the SoC group | At Month 3, Month 6 and Month 9
  To evaluate the effectiveness of inclisiran on the change in LDL-C levels at Month 3, Month 6, and Month 9, compared with SoC
The proportion of participants with LDL-C <1.8 mmol/L at 12 months, for the inclisiran group versus the SoC group | 12 months
  To evaluate the effectiveness of inclisiran on LDL-C at goal at Month 12
To describe LDL-C Test on Target value during the 12 months after baseline, for the inclisiran group and the SoC group. | 12 months
  To evaluate the real-world effectiveness of inclisiran, on LDL-C Test on Target at 1 year, compared with the SoC group.
The percentage change in levels of total cholesterol, triglyceride, HDL-C, Lp(a), ApoA, and ApoB, from baseline at 3 months, 6 months, 9 months, and 12 months, for the inclisiran group versus the SoC group | At Month 3, Month 6, Month 9, and Month 12
  To evaluate the effectiveness of inclisiran on the change in other parameters of the lipid profile at Month 3, Month 6, Month 9, and Month 12, compared with SoC
Area under the curve (AUC) of LDL-C level versus time (from 0 months to 12 months), for the inclisiran group versus the SoC group | Baseline, 12 months
  To evaluate the accumulated LDL-C in the inclisiran group and the SoC group
The proportion of participants with PDCinclisiran≥80% in the inclisiran group and the proportion of participants with PDCnon-statin≥80% in the SoC group, at 3 months, 6 months, 9 months, and 12 months | At Month 3, Month 6, Month 9, and Month 12
  To estimate the adherence to inclisiran and other non-statin lipid-lowering therapies (LLTs), as measured by the proportion of days covered (PDC), using prescription data
The average number of days covered, of inclisiran in the inclisiran group and of non-statin lipid-lowering therapies (LLTs) in the SoC group, at 3 months, 6 months, 9 months, and 12 months | At Month 3, Month 6, Month 9, and Month 12
  To estimate the adherence to inclisiran and other non-statin lipid-lowering therapies (LLTs), as measured by the proportion of days covered (PDC), using prescription data
The average PDCinclisiran in the inclisiran group and the average PDCnon-statin in the SoC group, at 3 months, 6 months, 9 months, and 12 months | At Month 3, Month 6, Month 9, and Month 12
  To estimate the adherence to inclisiran and other non-statin lipid-lowering therapies (LLTs), as measured by the proportion of days covered (PDC), using prescription data
Age at randomization and age at first diagnosis of CHD | 12 months
  To describe the demographics and clinical characteristics of the inclisiran group and the SoC group.
Sex | 12 months
  To describe the demographics and clinical characteristics of the inclisiran group and the SoC group
Temperature | 12 months
  To describe the demographics and clinical characteristics of the inclisiran group and the SoC group
Respiratory rate | 12 months
  To describe the vital signs characteristics of inclisiran group and the SoC group. It will be measured manually or with an electrocardiogram monitor.
Blood pressure | 12 months
  To describe the demographics and clinical characteristics of the inclisiran group and the SoC group
Heart rate | 12 months
  To describe the demographics and clinical characteristics of the inclisiran group and the SoC group
Previous lipid-lowering therapies (LLTs), through Adherence Assessment Questionnaire (AAQ) | 12 months
  The AAQ is a generic instrument for assessing non-adherence (NA) in chronic conditions, consists of 11 items in total. Ten of these items are phrased as statements and use a 4-point Likert scale, offering the response options: Strongly agree, Generally agree, Generally disagree, and Strongly disagree. Each item is scored from 1 to 4, with a higher score indicating a greater likelihood of non-adherence.
Previous lipid-lowering therapies (LLTs), through Adherence Barriers Questionnaire (ABQ) | 12 months
  The ABQ consists of 16 items, each addressing a specific adherence barrier. All items are formulated as statements. A 4-point Likert scale is used, deliberately omitting a neutral response option to encourage decisive answers. The available response options are: Strongly agree, Generally agree, Generally disagree, and Strongly disagree. Each response is assigned a value from 1 to 4 or 4 to 1, depending on the wording of the item, ensuring that a higher score reflects a stronger influence of a specific barrier on the patient's perception. The total score ranges from 16 (minimum) to 64 (maximum).Based on patient responses, both a general ABQ score and item- or subscale-specific scores can be calculated, indicating the number and strength of adherence barriers experienced by a patient.
Dose, frequency, and treatment duration of inclisiran in the inclisiran group and of other LLTs in the SoC group | 12 months
  To describe the treatment patterns of inclisiran and other LLTs
LDL-C variability in the inclisiran group by average successive variability (ASV), coefficient of variation (CV), and variation independent of mean (VIM) | 12 months
  To evaluate LDL-C variability in the inclisiran group
Subsequent LLTs for participants who discontinued/switched the assigned treatment | 12 months
  To describe the treatment patterns of inclisiran and other LLTs
Concomitant lipid lowering treatments | 12 months
  To describe the treatment patterns of inclisiran and other LLTs
Treatment satisfaction from Treatment Satisfaction Questionnaire for Medication (TSQM) | At Month 6 and Month 12
  This scale includes four dimensions: drug treatment effectiveness, adverse reactions, convenience, and overall satisfaction. Whether the patient has experienced adverse drug reactions is scored using "yes" and "no"; The adverse reaction dimension is evaluated using a Likert-5 scale, with scores ranging from 1 to 5 indicating "extremely dissatisfied" to "not dissatisfied at all"; The effectiveness, convenience, and overall satisfaction are rated on a Likert-7 scale, with scores ranging from 1 to 7 indicating "extremely dissatisfied" and "extremely satisfied", respectively. The standard score for each dimension is 100 points, and the higher the score, the higher the patient's satisfaction with drug treatment.
The average PDCinclisiran in the inclisiran group and the average PDCnon-statin in the SoC group, from patient questionnaire data, at 3 months, 6 months, 9 months, and 12 months | At Month 3, Month 6, Month 9, and Month 12
  To assess treatment satisfaction and adherence by questionnaires
Incidence of adverse events (AEs), serious adverse events (SAEs) | 12 months
  To evaluate the safety of Inclisiran
Number of participants with relevant medical history | 12 months
  To describe the demographics and clinical characteristics of the inclisiran group and the SoC group

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- China (18):
  - Novartis Investigative Site, Anqing, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Longyan, Fujian
  - Novartis Investigative Site, Jiamusi, Heilongjiang
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jining, Shandong
  - Novartis Investigative Site, Weifang, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigated Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang Uygur Autonomous Region
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Jinhua, Zhejiang
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.